CLINICAL TRIAL: NCT03215056
Title: A Randomised, Double-blind, Multicentre, Placebo Controlled Study to Evaluate the Safety and Efficacy of Methoxyflurane (PENTHROX®) for the Treatment of Acute Pain in Children and Adolescents from 6 to Less Than 18 Years of Age (presenting to an Emergency Department with Minor Trauma)
Brief Title: Methoxyflurane Analgesia for Paediatric Injuries
Acronym: MAGPIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Developments International Limited (Industry)
Collaborators: Pediatric Emergency Research in the UK and Ireland (PERUKI) (Other); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEOF-002; 2016-004290-41 (EudraCT Number)
Record Dates: First submitted 2017-07-02; First posted 2017-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENTHROX® (methoxyflurane) (Experimental): PENTHROX® (methoxyflurane) administered as a liquid for inhalation and should be self-administered under supervision of research nurse trained in its administration, using the hand held PENTHROX® inhaler.
  One vial of 3 mL PENTHROX® is to be vaporised in a PENTHROX® inhaler. On finishing the 3 mL dose, another 3 mL may be used.
  Dose of PENTHROX® should not exceed 6 mL in a single administration.
  The patient is instructed to inhale ten successive inhalations of PENTHROX® (methoxyflurane) followed by additional intermittent inhalations as required.
  The maximum dose administered will not exceed 6 mL of methoxyflurane.
  Interventions: Drug: Methoxyflurane
- Normal saline (Placebo Comparator): Normal saline will be administered as a liquid for inhalation and should be self-administered under supervision of research nurse trained in its administration, using the hand held PENTHROX® inhaler.
  One vial of 5 mL of normal saline is to be vaporised in a PENTHROX® inhaler. On finishing the 5 mL dose, another 5 mL may be used.
  Dose of normal saline should not exceed 10 mL in a single administration.
  In this study, the patient is instructed to inhale ten successive inhalations of placebo followed by additional intermittent inhalations as required.
  The maximum dose administered will not exceed 10 mL of placebo (2 × 5 mL)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Methoxyflurane — PENTHROX 3mL inhalation vapour, liquid
  Other Names: Penthrox®
  Arms: PENTHROX® (methoxyflurane)
Drug: Normal saline — Placebo
  Arms: Normal saline

SUMMARY:
This is a randomised, double-blind, multicentre, placebo controlled study to evaluate the safety and efficacy of methoxyflurane (Penthrox®) for the treatment of acute pain in children and adolescents from 6 to less than 18 years of age (presenting to an Emergency Department with minor trauma). It is conducted as part of the Paediatric Investigation Plan (PIP) agreed with the Paediatric Committee (PDCO) of the European Medicines Agency (EMA).

The study aims to provide evidence under blinded controlled conditions that Penthrox is safe and effective in patients aged 6 to less than 18 years presenting to ED with pain associated with minor trauma.

DETAILED DESCRIPTION:
This is a randomised, double-blind, multicentre, placebo-controlled study in children and adolescents aged 6 to less than 18 years presenting to an ED requiring analgesia for acute pain, with visual analogue scale (VAS) score of 55 to 85 mm or Wong-Baker Faces score of 6 to 8 associated with minor trauma. In the context of the current study, minor trauma refers to "a non-critical and non-limb threatening physical wound or injury of the tissues", such as, soft tissue injuries, fractures of the extremities, burns, penetration by foreign bodies, lacerations, dislocation, contusions, etc.

This study will include screening and enrolment, followed by treatment and day 14 ± 2 day safety follow-up post treatment. The procedure for screening and enrolment including obtaining consent/assent is to occur on the same day. The expected duration for each patient in the study is up to 16 days.

The clinician/research nurse must ascertain that the patient has not been pre-medicated with an analgesic within 5 hours prior to randomisation, except Entonox (50% nitrous oxide and 50% oxygen mixture) which is prohibited within 30 minutes prior to randomisation, diclofenac which is prohibited within 8 hours prior to randomisation or oral morphine which is prohibited within 10 hours prior to randomisation.

At least 220 eligible children and adolescents aged 9 to < 18 years (110 children aged 9 to < 12 years and 110 adolescents aged 12 to < 18 years) were to be randomised in a 1:1 ratio to receive either methoxyflurane or placebo from the PENTHROX inhaler. Additionally, at least 36 eligible children aged 6 to < 9 years were to be randomized in a 1:1 ratio. Randomisation was stratified by age group (6 to < 9 years; 9 to < 12 years; 12 to < 18 years).

Pain scores will be assessed using the VAS or Wong-Baker FACES® Pain Rating scale in younger children who cannot utilise the VAS tool. A pain score will be measured at screening to establish study eligibility. After randomisation, a baseline pain score will be recorded between 5 to 60 minutes after the screening pain score and will act as a validation score. If the baseline pain score falls outside the range of 55 to 85 mm on the VAS or 6 to 8 on Wong-Baker FACES Pain Rating scale, the patient will be withdrawn from the study (randomised, but not treated). Patients who have a pain score between 55 and 85 mm on the VAS or 6 to 8 on Wong-Baker FACES Pain Rating scale at screening and baseline will be eligible to receive treatment. In order to improve patient recruitment, a protocol amendment in July 2019 widened the range of the eligible VAS pain score from 60 to 80 mm to 55 to 85 mm. However, this amendment was quite late in study conduct and shortly prior to the COVID pandemic, hence the majority of patients were recruited under the original criterion (60 to 80mm).

Following enrolment and initial assessments, the research nurse will assist the patient to self administer ten successive inhalations of PENTHROX® (methoxyflurane) or placebo. The research nurse, the treating clinician and the patient will be blind to the treatment administered.

Patients/parents/legal guardians will be advised that rescue medication will be available immediately on request at any time during or after the completion of the treatment. The rescue medication to be used will be at the discretion of the blinded clinician. Rescue analgesia should be near the potency equivalence of active PENTHROX. Depending on the standard practice of the participating site, this may include intranasal fentanyl, intranasal diamorphine, intranasal ketamine, Entonox (50% nitrous oxide and 50% oxygen mixture), intravenous morphine, or oral morphine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6 to less than 18 years.
2. Attending ED following minor trauma.
3. Evidence of signed and dated informed consent/assent document indicating that the patient (and/or a parent/legal guardian) has been informed of all pertinent aspects of the study*.
4. Pain scores 55 to 85 mm as measured using VAS or 6 to 8 using Wong-Baker FACES Pain Rating scale.

Note: the range for VAS pain scores was widened from 60 to 80 mm to 55 to 85 mm to improve patient recruitment but very few patients were recruited after that amendment.

Exclusion Criteria:

1. Critical, life-or limb-threatening condition requiring immediate management.
2. Open fractures.
3. Patients with any other clinical condition that may, in the opinion of the Investigator, impact the patient's ability to participate in the study, or the study results.
4. Patients deemed not cognitively capable of effectively self-administering the study drug using the PENTHROX® inhaler.
5. Treatment with any analgesic agent within 5 hours prior to randomisation, except Entonox (50% nitrous oxide and 50% oxygen mixture) which is prohibited within 30 minutes prior to randomisation, diclofenac which is prohibited within 8 hours prior to randomisation or oral morphine which is prohibited within 10 hours prior to randomisation.
6. Patients with chronic pain.
7. Patients having received an Investigational Medicinal Product (IMP) in the preceding 3 months.
8. Known pregnancy or breastfeeding females.
9. Personal or familial hypersensitivity to PENTHROX® or any fluorinated anaesthetics.
10. Patients requiring oxygen therapy.
11. Patients with known or genetic susceptibility to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives.
12. Clinically evident respiratory depression.
13. Previous use of methoxyflurane (including as an IMP).
14. History of signs of liver damage including after previous PENTHROX® (methoxyflurane) use or halogenated hydrocarbon anaesthesia.
15. Known significant renal impairment.
16. Altered level of consciousness due to any cause including head injury, drugs, or alcohol.
17. Known significant cardiovascular instability (e.g., pathological arrhythmia).
18. Inability to participate in telephonic follow-up on (Day 14 ± 2 days) as per study requirement

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity between methoxyflurane and placebo as measured by change from baseline in VAS pain scores at 15 minutes for patients aged 9 to < 18 years. | Baseline to 15 minutes
  The primary analysis was conducted using an analysis of covariance (ANCOVA) model with change from baseline in pain score at 15 minutes as the dependent variable, continuous baseline pain, treatment and age group (9 to < 12 years versus 12 to < 18 years) as fixed effects and centre (site) as a random effect. Missing pain scores at 15 (± 2) minutes were imputed using worst observation carried forward (WOCF) and pain scores taken after the initiation of rescue medication were included.
  Note the population for the primary analysis was changed in the protocol following an amendment to the sample size across the age groups due to difficulties recruiting patients into the youngest (6 to < 9 years) age group and agreement with agencies to focus the primary analysis on 9 to < 18-year-olds.

SECONDARY OUTCOMES:
Difference in pain intensity between methoxyflurane and placebo as measured by change from baseline in VAS pain scores at 15 minutes in the ITT Population (patients aged 6 to <18 years). | Baseline to 15 minutes
  This analysis used the same statistical model (ANCOVA) as the primary analysis.
Responder analysis - number of responders, who achieve 30% reduction in VAS score compared to baseline, at 15 minutes in the ITT population (patients aged 6 to <18 years). | Baseline to 15 minutes
  Patients with missing data at baseline or 15 minutes were regarded as non-responders. Data were analysed using a logistic regression model adjusted for continuous baseline pain score, age group and treatment. Number and percentage of responders are presented for each treatment group. Treatment effect is presented as the OR with the corresponding 95% CI and p-value.
Longitudinal analysis of VAS pain scores at 5, 10, 15, and 20 minutes following commencement of treatment in the ITT population (patients aged 6 to <18 years). | Baseline to 5, 10, 15 and 20 minutes
  Data were analysed using a mixed model repeated measure (MMRM) approach with age group, continuous baseline pain score, assessment time (5, 10, 15 and 20 minutes), treatment group, and assessment time by treatment group interaction.
Number of inhalations taken before first pain relief is summarised by category (1 to 10 inhalations, 11 to 20 inhalations, 21 to 30 inhalations, >30 inhalations, or no relief recorded) in the ITT population (patients aged 6 to <18 years). | From baseline until time at which first pain relief is reported, assessed up to Emergency Department discharge or inpatient admission.
  Additionally, for patients with pain relief documented prior to discharge, continuous descriptive summaries are presented for the number of inhalations.
Rescue medication requested within 20 (+2 minutes) minutes of start of treatment and any time during treatment in the ITT population (patients aged 6 to <18 years). | From baseline until request of rescue medication, assessed until point of either Emergency Department discharge or inpatient admission.
  These endpoints were analysed using a logistic regression model as described for the pain responder analysis.
The time to request for rescue medication in the ITT population (patients aged 6 to <18 years). | From baseline until time at which rescue medication is first requested, assessed up to time of Emergency Department discharge or inpatient admission.
  Patients who did not receive rescue medication were censored. Data was analysed using a Cox proportional hazards model stratified by age group and adjusted for treatment and continuous baseline VAS score to obtain an estimate of the hazard ratio (methoxyflurane/placebo) and the corresponding two-sided 95% CI. The p-value was obtained from a stratified log-rank test (stratified by age group).
The time to first pain relief derived as time in minutes since start of study treatment until first pain relief in the ITT population (patients aged 6 to <18 years). | From baseline until time at which first pain relief is reported, assessed up to Emergency Department discharge or inpatient admission.
  Patients who did not experience pain relief by the time of discharge were censored at their time of discharge (or last VAS assessment date if date of discharge is missing). This endpoint was analysed using a Cox PH model as described above for time (minutes) to request rescue medication.
Number of inhalations taken before first pain relief split by whether the hole was covered at least once or not covered in the ITT population (patients aged 6 to <18 years). | Baseline until time at which first pain relief is reported, assessed up to Emergency Department discharge or inpatient admission..
  Data was summarised using the same categories as for number of inhalations taken before first pain relief split by dilutor hole covered at least once/not covered.
Global medication performance assessment by patient, clinician and research nurse: 0 = poor to 4 = excellent, measured after completion of treatment. | From baseline, assessed up to Emergency Department discharge or inpatient admission.
  An ordinal logistic regression was performed with adjustments for continuous baseline pain score, age group and treatment. Number and percentage of patients per response score per treatment group are presented. Treatment effect is presented as the OR with the corresponding 95% CI and p-value (obtained using profile likelihood).
Heart rate | From baseline to 5, 10, 15, 20 and 30 minutes, followed by a 30-minute interval thereafter assessed until the point of either Emergency Department discharge or inpatient admission.
  Absolute and change from baseline in heart rate [bpm], at each scheduled protocol timepoint, were listed and plotted (boxplots) by scheduled protocol timepoint.
Respiratory rate | From baseline to 5, 10, 15, 20 and 30 minutes, followed by a 30-minute interval thereafter assessed until the point of either Emergency Department discharge or inpatient admission.
  Absolute and change from baseline in respiratory rate [breaths/min] at each scheduled protocol timepoint, were listed and plotted (boxplots) by scheduled protocol timepoint.
Oxygen saturation | From baseline to 5, 10, 15, 20 and 30 minutes, followed by a 30-minute interval thereafter assessed until the point of either Emergency Department discharge or inpatient admission.
  Absolute and change from baseline in oxygen saturation [%] at each scheduled protocol timepoint, were listed and plotted (boxplots) by scheduled protocol timepoint.

OTHER OUTCOMES:
Treatment-emergent adverse events (TEAEs); all, prior to discharge and post discharge up to (14 ± 2 days following ED discharge/inpatient decision). | Baseline until 14 days post discharge
  The safety outcome variables will be analysed by means of descriptive statistics. All TEAEs (including the safety follow up period) are reported with some tables repeated for TEAEs recorded prior to discharge and TEAEs recorded post discharge (as part of the 14-day safety follow up call).
Patient sedation score based on University of Michigan Sedation Scale (UMSS). | Baseline to 5, 10, 15, 20 and 30 minutes, followed by a 30-minute interval thereafter, assessed up to ED discharge/inpatient admission.
  The UMSS assesses the level of alertness on a 5-point scale ranging from score 0 (awake and alert) to score 4 (unarousable). A shift table presents baseline scores versus worst score during study treatment. Baseline versus discharge scores are also presented.
Blood pressure | From baseline to 5, 10, 15, 20 and 30 minutes, followed by a 30-minute interval thereafter assessed until the point of either Emergency Department discharge or inpatient admission.
  Absolute and change from baseline in systolic blood pressure [mmHg] and diastolic blood pressure [mmHg], at each scheduled protocol timepoint, were listed and plotted (boxplots) by scheduled protocol timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Hartshorn, Principal Investigator — Birmingham Children's Hospital
Locations (11):
- Our Lady's Children's Hospital, Crumlin, Dublin, Ireland
- United Kingdom (10):
  - Royal Aberdeen Children's Hospital, Aberdeen, Aberdeenshire
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Royal Alexandra Children's Hospital, Brighton, East Sussex
  - Royal London Hospital, London, Greater London
  - Alder Hey Children's Hospital, Liverpool, Merseyside
  - Nottingham University Hospitals City Campus, Nottingham, Notttinghamshire
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - Leicester Royal Infirmary, Leicester
  - Ormskirk District Hospital, Ormskirk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartshorn S, Barrett MJ, Lyttle MD, Yee SA, Irvine AT; in collaboration with Paediatric Emergency Research in the UK and Ireland (PERUKI). Inhaled methoxyflurane (Penthrox(R)) versus placebo for injury-associated analgesia in children-the MAGPIE trial (MEOF-002): study protocol for a randomised controlled trial. Trials. 2019 Jul 4;20(1):393. doi: 10.1186/s13063-019-3511-4. PMID 31272493
- [Derived] Hartshorn S, Barrett MJ, Bloom B, Lyttle MD, Walton E, Steel K, Yee SA, Irvine A; Paediatric Emergency Research in the United Kingdom & Ireland (PERUKI). Treatment of acute trauma-related pain in children and adolescents with methoxyflurane (Penthrox(R)) compared to placebo (MAGPIE): A randomised clinical trial. Injury. 2025 Dec;56(12):112830. doi: 10.1016/j.injury.2025.112830. Epub 2025 Oct 20. PMID 41242203